CLINICAL TRIAL: NCT04671602
Title: Implementing LEANBH Ambulatory Integrated Blood Pressure Monitoring in Maternity Services
Brief Title: Learning to Evaluate Blood Pressure at Home (LEANBH)
Acronym: LEANBH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College Cork (Other)
Collaborators: Science Foundation Ireland (Other)
Responsible Party: Principal Investigator, Fergus McCarthy, Consultant Obstetrician, University College Cork
Other Study IDs: FMC01UCC2020
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hypertension in Pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 has highlighted important deficiencies in our health service where front line staff and pregnant women are being exposed to SARS-Cov-2 through assessments that could be conducted using Connected Health solutions, reducing risks of contracting or disseminating SARS-Cov-2. Currently, pregnant women are not attending GPs or hospitals for BP monitoring for fear of contracting SARS-Cov-2. Uncontrolled or unmonitored hypertension in pregnancy is associated with maternal and fetal morbidity and mortality. The aim of the study is to use home BP monitoring as an adjunct to standard care for women with borderline/suspected hypertension in pregnancy. To reduce the exposure risk for staff and pregnant women, we propose the immediate implementation of ambulatory automated self BP monitoring using the LEANBH platform- an existing integrated platform to monitor pregnant women.

DETAILED DESCRIPTION:
The COVID-19 pandemic exposes our front-line staff to unnecessary risks in interacting with COVID-19 affected patients. Current care of pregnant women who have uncontrolled/unmonitored hypertension involves multiple visits to obstetric units for blood pressure checks. These visits put the women at risk of contracting or transmitting SARS-CoV-2 by bringing them into hospitals for checks which could otherwise be done remotely. Up to 20% of pregnant women will experience a hypertensive episode during pregnancy or the postpartum period. Uncontrolled or unmonitored hypertension in pregnancy may be associated with significant maternal and fetal morbidity and mortality including pre-eclampsia, stroke and stillbirth. The current management of suspected hypertension in pregnancy involves prolonged admission to hospital for BP monitoring or multiple visits to day assessment units or primary care physicians. All of these increase the risk of contracting or transmitting SARS-CoV-2. In addition, pregnant women with COVID-19 who are receiving inpatient care also require regular BP monitoring increasing the exposure risk for staff of contracting SARS-CoV-2. Pregnant women not attending GPs or hospitals for BP monitoring out of fear of contracting COVID-19 drastically increase their risk of suffering adverse effects from undiagnosed or uncontrolled hypertension. The ideal solution would be to facilitate inpatient or outpatient monitoring with reduced face to face contact between staff and infected patients. This would ensure a safer experience for all by reducing the risk of contracting SARS-CoV-2 while safely offering remote BP monitoring. LEANBH offers this safe alternative to direct hospital contact for pregnant women and staff by providing ambulatory automated self BP monitoring using the LEANBH integrated platform. This proposal will deliver immediate ambulatory BP self-monitoring performed remotely without need for direct physical contact, minimising risk of exposure to SARS-CoV-2 for staff and pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over.
* Ability to give informed consent.
* Mobile application compatible smartphone.
* Increased requirement for blood pressure monitoring in this pregnancy as determined by their treating obstetric team.
* Between 12 weeks of pregnancy and up to six weeks postpartum

Exclusion Criteria:

* Inability to give informed consent (language barrier)
* Confirmed Preeclampsia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All legally adult women with an ongoing, confirmed intrauterine pregnancy.
Study Population: Women with an ongoing, confirmed intrauterine pregnancy who have borderline high blood pressure or are at risk of developing high blood pressure in this pregnancy and are due to give birth in Cork University Maternity Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Participant Satisfaction | 12-42 weeks gestation
  The primary outcome measure will be participant satisfaction with home blood pressure monitoring. Once a participant completes the LEANBH Study, an online system usability scale will be sent to all participants. This questionnaire contains 35 questions which will accurately capture user experience and satisfaction while participating in the study.

SECONDARY OUTCOMES:
Clinical Escalation | 12-42 weeks gestation
  The secondary outcome measure is the clinical escalation offered to participants as part of the LEANBH study. Home BP readings will be reviewed daily and clinical escalation offered when appropriate throughout the study.
Adverse Events | 12 weeks gestation - 6 weeks postpartum
  Preeclampsia, Preterm Delivery, IUGR, Postnatal Hospital Stay and Admission to NNU will all be considered as adverse events for the purpose of this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Cork University Maternity Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No